CLINICAL TRIAL: NCT02842008
Title: Effects of a Therapeutic Exercise Program for Injuries Prevention in Wheelchair Basketball (WB) Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Saleky García Gómez, PT PhD student, Universidad Politecnica de Madrid
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UPMadrid
Record Dates: First submitted 2016-06-06; First posted 2016-07-22 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Athletic Injuries; Shoulder Pain; Shoulder Injury
Keywords: Exercise Therapy; Shoulder pain; Shoulder injuries; Shoulder function; Prevention; Wheelchair users
MeSH Terms: conditions — Athletic Injuries; Shoulder Pain; Shoulder Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): Wheelchair basketball players participating in home therapeutic exercise program that use the protocol of postural hygiene.
  Interventions: Behavioral: Exercise group
- Control group (No Intervention): Wheelchair basketball players that not participate in home therapeutic exercise program and use a protocol of postural hygiene provided.

INTERVENTIONS:
Behavioral: Exercise group — This group will receive a home exercise program of shoulder based on mobility, strength and strengthening exercises, lasting 10 weeks, 3 times per weeks. The target dose use for mobility consisted in 8 repetitions for each 4 movements, for strengthening using resistive bands, 3 sets (including 5 exercises) of 10 repetitions with a 45 second rest between sets and 5 repetitions for each 5 strength with a 30 second rest and general protocol of postural hygiene. The instructional of the program is 30 minutes each day during the time of the study (10 weeks) with a screening about the exercise program and the daily activities performed every 4 weeks. Physiotherapist provided support to subjects through email along 10 weeks.
  Arms: Exercise group

SUMMARY:
Shoulder pain is the most common symptom of physical dysfunction in wheelchair basketball players. About the 85% of this population had shoulder pain in some moment of their life. Some studies suggest that exercise is an important tool as an element to treat and prevent shoulder injuries. For that reason, an intervention program would be a useful tool for prevent shoulder injuries in this population.

The purpose of this study is determine the effects of therapeutic exercise program wheelchair basketball players, in order to prevent shoulder injuries.

DETAILED DESCRIPTION:
The hypothesis of the study was that the exercise program was effective to prevent shoulder injuries in this population.

ELIGIBILITY:
Study Population 36 wheelchair basketball players belonging to the male and female preselection Spanish wheelchair basketball national team were recruiting during a campus. The inclusion and exclusion criteria were chosen to include a specific population.

Inclusion Criteria:

* Players belonging to the male and female preselection Spanish wheelchair basketball national team.
* Have the federal license at the Spanish Sport Federation for People with Physical Disabilities available at the time of the study (2015-2016 season).
* For players using wheelchair for daily activities, to use the manual wheelchair at least for 3 hours a day and 6 hours of wheelchair basketball training per week.
* For players not using wheelchair for daily activities, to use the manual wheelchair at least for 6 hours of wheelchair basketball training per week.
* Use wheelchair at least one year before the study and at least one year of experience in the sport competition.
* Acceptance of informed consent.

Exclusion Criteria:

* History of acute injuries in the post-surgical process or dislocation along the year before the study. These conditions may affect the effective of the exercise intervention.
* Differential diagnosis as acute injuries at cervical region and recent traumatic injury in shoulder one year before the study. The exercise program may not be appropriate for these conditions.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline shoulder pain at 10 weeks | Baseline and at 10 weeks
  The presence of shoulder pain will be measured at the beginning and at 10 weeks with "Shoulder Pain Index for Wheelchair Basketball (SPI-WB)" (submitting).

SECONDARY OUTCOMES:
Neer test | Baseline and at 10 weeks
  Neer's Test assesses for possible rotator cuff impingement. Pain is a positive test.
Hawkins-Kennedy test | Baseline and at 10 weeks
  Hawkins-Kennedy's test indicative a possible impingement between the greater tuberosity of the humerus against the coraco- humeral ligament.
Jobe test | Baseline and at 10 weeks
  Jobe's test assesses for possible supraspinatus weakness and/or impingement.
Patte test | Baseline and at 10 weeks
  Patte's test measure for possible infraspinatus and teres minor weakness and/or impingement.
Shoulder range of motion | Baseline and at 10 weeks
  The range of motion will be evaluated in flexion, extension, internal rotation, external rotation and abduction with a goniometric at the beginning and at 10 weeks.
Players´ adherence to the exercise program | At 4 and 8 weeks
  Players will complete a questionnaire rating their adherence to the exercise program.
Players´ self-efficacy to the exercise program | Baseline
  Players will complete a questionnaire about the self-efficacy according to the exercise program.
Players adherence to the protocol of postural hygiene. | At 4 and 8 weeks
  Players will complete a follow-up questionnaire rating their adherence to the protocol of postural hygiene.
Activities performed outside of the training and exercise program. | At 4 and 8 weeks
  Players will be complete a follow-up questionnaire about the activities performed outside of the training and exercise program.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Pérez Tejero, PhD, Study Director — Universidad Politecnica de Madrid
Locations (1):
- Universidad Politécnica de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided